CLINICAL TRIAL: NCT04833790
Title: What Drives Poor Care for Child Diarrhea: A Standardized Patient Experiment
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RAND (Other)
Responsible Party: Principal Investigator, Zachary Wagner, Professor of Policy Analysis, RAND
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 1R01DK126049-01A1 (NIH)
Record Dates: First submitted 2021-04-02; First posted 2021-04-06 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Child Diarrhea

STUDY DESIGN:
Intervention Model Description: The two interventions are patient type (4 types) and free distribution of treatment for child diarrhea (2 groups). These will be cross-randomized creating 8 study arms.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The study participants are private health care providers in India who treat child diarrhea. Providers will be masked to which type of patient they are assigned to but not whether they receive free treatment for child diarrhea. Outcomes will assessed by anonymous standardized patients and these will be blind to whether the provider received free treatment for child diarrhea.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Free distribution of ORS + standardized patient with ORS preference (Experimental): Providers assigned to this arm will receive 3 months supply of ORS. Roughly 4 weeks later, they will receive a visit from a standardized patient (outcomes assessor) who poses as a caretaker for their child with diarrhea and indicates a preference for ORS.
  Interventions: Behavioral: Free distribution of ORS; Behavioral: Standardized patient with ORS preference
- Free distribution of ORS + standardized patient with Antibiotic preference (Experimental): Providers assigned to this arm will receive 3 months supply of ORS. Roughly 4 weeks later, they will receive a visit from a standardized patient (outcomes assessor) who poses as a caretaker for their child with diarrhea and indicates a preference for Antibiotics.
  Interventions: Behavioral: Free distribution of ORS; Behavioral: Standardized patient with Antibiotic preference
- Free distribution of ORS + standardized patient with no preference (Experimental): Providers assigned to this arm will receive 3 months supply of ORS. Roughly 4 weeks later, they will receive a visit from a standardized patient (outcomes assessor) who poses as a caretaker for their child with diarrhea and indicates no preference for treatment.
  Interventions: Behavioral: Free distribution of ORS; Behavioral: Standardized patient with no preference
- Free distribution of ORS + standardized patient with no preference + no financial incentive (Experimental): Providers assigned to this arm will receive 3 months supply of ORS. Roughly 4 weeks later, they will receive a visit from a standardized patient (outcomes assessor) who poses as a caretaker for their child with diarrhea and indicates no preference for treatment and indicates that they will purchase whatever the provider recommends from a relative's drug shop.
  Interventions: Behavioral: Free distribution of ORS; Behavioral: Standardized patient with no preference + no financial incentive
- Status quo ORS supply + standardized patient with ORS preference (Experimental): Providers assigned to this arm will have status who ORS supply. Roughly 4 weeks later, they will receive a visit from a standardized patient (outcomes assessor) who poses as a caretaker for their child with diarrhea and indicates a preference for ORS.
  Interventions: Behavioral: Standardized patient with ORS preference
- Status quo ORS supply + standardized patient with Antibiotic preference (Experimental): Providers assigned to this arm will have status who ORS supply. Roughly 4 weeks later, they will receive a visit from a standardized patient (outcomes assessor) who poses as a caretaker for their child with diarrhea and indicates a preference for Antibiotics.
  Interventions: Behavioral: Standardized patient with Antibiotic preference
- Status quo ORS supply + standardized patient with no preference (Experimental): Providers assigned to this arm will have status who ORS supply. Roughly 4 weeks later, they will receive a visit from a standardized patient (outcomes assessor) who poses as a caretaker for their child with diarrhea and indicates no preference for treatment.
  Interventions: Behavioral: Standardized patient with no preference
- Status quo ORS supply + standardized patient with no preference + no financial incentive (Experimental): Providers assigned to this arm will have status who ORS supply. Roughly 4 weeks later, they will receive a visit from a standardized patient (outcomes assessor) who poses as a caretaker for their child with diarrhea and indicates no preference for treatment and indicates that they will purchase whatever the provider recommends from a relative's drug shop.
  Interventions: Behavioral: Standardized patient with no preference + no financial incentive

INTERVENTIONS:
Behavioral: Free distribution of ORS — Provides will receive 3 months supply of ORS at the beginning of the study to dispense to their patients. They will be asked to dispense the ORS at the market rate and not to give it away to other providers.
  Arms: Free distribution of ORS + standardized patient with Antibiotic preference; Free distribution of ORS + standardized patient with ORS preference; Free distribution of ORS + standardized patient with no preference; Free distribution of ORS + standardized patient with no preference + no financial incentive
Behavioral: Standardized patient with ORS preference — Providers will receive a visit from an anonymous standardize patient posing a caretaker for a child with diarrhea who requests ORS to treat their child's diarrhea.
  Arms: Free distribution of ORS + standardized patient with ORS preference; Status quo ORS supply + standardized patient with ORS preference
Behavioral: Standardized patient with Antibiotic preference — Providers will receive a visit from an anonymous standardize patient posing a caretaker for a child with diarrhea who requests Antibiotics to treat their child's diarrhea.
  Arms: Free distribution of ORS + standardized patient with Antibiotic preference; Status quo ORS supply + standardized patient with Antibiotic preference
Behavioral: Standardized patient with no preference — Providers will receive a visit from an anonymous standardize patient posing a caretaker for a child with diarrhea who does not request anything specific to treat their child's diarrhea.
  Arms: Free distribution of ORS + standardized patient with no preference; Status quo ORS supply + standardized patient with no preference
Behavioral: Standardized patient with no preference + no financial incentive — Providers will receive a visit from an anonymous standardize patient posing a caretaker for a child with diarrhea who does not request anything specific to treat their child's diarrhea. In addition they will inform the provider that they are not going to purchase anything from the provider because they have an uncle with a drug shop where they can get a discount.
  Arms: Free distribution of ORS + standardized patient with no preference + no financial incentive; Status quo ORS supply + standardized patient with no preference + no financial incentive

SUMMARY:
Diarrhea is the second leading cause of death for children around the world, although nearly all of these deaths could be prevented with an inexpensive and simple treatment: oral rehydration salts (ORS). Many children with diarrhea do not receive ORS when they seek treatment and this study uses a field experiment to examine why this occurs. We will use anonymous standardized patients combined with a randomized ORS supply intervention to isolate the causal effect of several potential reasons for why children do not receive ORS when they seek care: 1) caretakers prefer ORS alternatives, 2) providers have a financial incentives to prescribe ORS alternatives, and 3) ORS is often out of stock.

DETAILED DESCRIPTION:
Diarrhea is the second leading cause of death for children around the world. This is true despite the fact that nearly all such deaths could be prevented with a simple and inexpensive solution: oral rehydration salts (ORS). Private health care providers, who treat the majority of childhood illness in low- and middle-income countries (LMICs), are particularly unlikely to dispense ORS to children with diarrhea. Instead, providers often dispense antibiotics inappropriately. Recognizing this significant challenge, several international organizations (including USAID) have invested heavily in trying to increase ORS dispensing in the private sector. In the absence of evidence on why ORS is so inconsistently dispensed by private providers, however, several interventions to promote private sector ORS dispensing have been ineffective. Clearly, a critical and urgent next step is to examine the key drivers of underprescription of ORS and overprescription of antibiotics in the private sector in order to inform efforts to improve diarrhea care. In this study, we examine several leading explanations for poor quality of care for child diarrhea in the private sector. First, patient preferences for ORS alternatives (e.g., an antibiotic) could be driving underprescription of ORS. We will identify the causal effect of patient preferences (Aim 1) by having anonymous standardized patients (SPs) pose as caretakers of children with diarrhea and express different (randomly assigned) preferences for treatment (ask for ORS, ask for antibiotics, or let provider decide). Second, private providers could be responding to financial incentives to sell more profitable alternatives to ORS (e.g., an antibiotic). To estimate the causal effect of financial incentives (Aim 2), we will instruct a subset of SPs to inform providers that they can get discounted treatments at a relative's drug shop. This eliminates the provider's financial incentive to recommend a given treatment and allows us to estimate the effect of such incentives. Finally, private providers might not directly distribute ORS or could have frequent stock-outs. To estimate the causal effect of stock-outs (Aim 3), we will randomly assign half of the providers to receive a three-month supply of ORS. This generates exogenous variation in stock outs and thus enables us to isolate the causal effect of stock outs on ORS and antibiotic prescribing. Combining, (a) causal estimates of the impact of each factor on prescribing, and (b) population estimates of the prevalence of each factor, will allow us to estimate the population level impact of implementing interventions that address each factor (Aim 4). This study will provide the most comprehensive evidence to date on why one of the most important health technologies in history is often not prescribed. The results will inform the design of interventions aimed at increasing ORS dispensing and reducing antibiotic dispensing. If such interventions are targeted appropriately, millions of young lives could be saved.

ELIGIBILITY:
Inclusion Criteria:

* Eligible providers will be private providers over 18 years old in our sampled villages that treat at least one case of child diarrhea per week

Exclusion Criteria:

* Providers in villages where there are no other providers will be excluded for confidentiality concerns

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2451 (Actual)
Dates: Start 2022-05-05 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Received or prescribed ORS | 4 weeks after the ORS supply is dispensed. Same time as standardize patient visits occur.
  Standardized patients will record whether the provider either dispensed or prescribed ORS for their child's diarrhea .
Received or prescribed antibiotic | 4 weeks after the ORS supply is dispensed. Same time as standardize patient visits occur.
  Standardized patients will record whether the provider either dispensed or prescribed antibiotics for their child's diarrhea.

SECONDARY OUTCOMES:
Received or prescribed zinc | 4 weeks after the ORS supply is dispensed. Same time as standardize patient visits occur.
  Standardized patients will record whether the provider either dispensed or prescribed zinc for their child's diarrhea.
Received or prescribed zinc+ORS | 4 weeks after the ORS supply is dispensed. Same time as standardize patient visits occur.
  Standardized patients will record whether the provider either dispensed or prescribed zinc and ORS (the gold standard treatment) for their child's diarrhea.
Received or prescribed ORS and no antibiotics | 4 weeks after the ORS supply is dispensed. Same time as standardize patient visits occur.
  Standardized patients will record whether the provider either dispensed or prescribed ORS and no antibiotics for their child's diarrhea.
Received or prescribed ORS + zinc and no antibiotics | 4 weeks after the ORS supply is dispensed. Same time as standardize patient visits occur.
  Standardized patients will record whether the provider either dispensed or prescribed ORS and zinc with no antibiotics for their child's diarrhea.

CONTACTS AND LOCATIONS:
Locations (1):
- Indian Institute of Management Bangalore, Bangalore, Karnataka, India

IPD SHARING:
Plan to Share IPD: Undecided
We plan on making individual underlying data available for replication purposes but this plan needs to be finalized with our IRB